CLINICAL TRIAL: NCT06339112
Title: The Effect of Playing With a Toy Nebulizer and Watching Cartoons on the Fear and Anxiety of 4-6-year-old Children Who Are Administered Inhaler Medication.
Brief Title: The Effect of Playing With a Toy Nebulizer and Watching Cartoons on the Fear and Anxiety on Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tarsus University (Other)
Responsible Party: Principal Investigator, Atiye Karakul, Assoc. Prof, Tarsus University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2024/10
Record Dates: First submitted 2024-03-24; First posted 2024-04-01 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Fear; Anxiety; Inhalant Use
Keywords: fear; anxiety; children; emergency
MeSH Terms: conditions — Anxiety Disorders; Emergencies

STUDY DESIGN:
Intervention Model Description: A randomized controlled experimental study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Playing with toy nebulizer (Experimental): The child who needs to take inhaler medication is taken to the observation room. Before starting the procedure, the child will be introduced to the toy nebulizer. The toy nebulizer is shown to the child as an example and allowed to play with it so that the level of fear can be reduced.
  Interventions: Other: Playing with toy nebulizer
- Cartoon (Experimental): Approximately 10 minutes for the child. Inhaler medication will be given with a mask that lasts. 2-3 minutes before starting drug treatment, the child will be allowed to watch cartoons according to his age group and will be encouraged to do so throughout the procedure. Vital signs (pulse, blood pressure, SPo2, respiration) before and after the application of the Child Fear Scale will be evaluated by the researcher and the parent and recorded in the intervention follow-up form by the researcher.
  Interventions: Other: Cartoon
- Control (No Intervention): Routine care will be provided.

INTERVENTIONS:
Other: Playing with toy nebulizer — The child who needs to take inhaler medication is taken to the observation room. Before starting the procedure, the toy nebulizer is introduced to the child. The toy nebulizer is shown to the child as an example and allowed to play, thus reducing the level of fear. Inhaler medication is given through a mask for 10 minutes. Vital signs (pulse) before and after the application. , blood pressure, SPo2, respiration), the Child Fear Scale will be evaluated by the researcher and the parent and recorded in the intervention follow-up form by the researcher.
  Arms: Playing with toy nebulizer
Other: Cartoon — Approximately 10 minutes for the child. Inhaler medication will be given with a mask that lasts. 2-3 minutes before starting drug treatment, the child will be allowed to watch cartoons according to his age group and will be encouraged to do so throughout the procedure.
  Vital signs (pulse, blood pressure, SPo2, respiration) before and after the application, the Child Fear Scale will be evaluated by the researcher and the parent and recorded in the intervention follow-up form by the researcher.
  Arms: Cartoon

SUMMARY:
This research was planned as a randomized controlled experimental type to determine the effect of playing with a toy nebulizer and watching cartoons on children's fear and physiological parameters in 3-6 year old children who were administered inhaler medication. The population of the study, planned as a randomized controlled experimental study, will consist of 4-6 year old children who apply to Tarsus State Hospital pediatric services and receive inhaler treatment. According to the power analysis performed for the sample size, the power of the sample was calculated with the G*Power 3.1 program, in line with the literature (Durak 2019; Özsamuri 2020). While the amount of Type I error was 0.05 and the power of the test was 0.95 (α= 0.05, 1-β= 0.95), the minimal sample size was calculated as 105 children (35 children in each group). Considering the possible losses from the sample for any reason during the study period, it was planned to increase the number of samples by 10% and include 38 children in the study and control groups. Child Information Form, Fear Assessment Scale and Child Anxiety Scale-State Scale will be used to collect data.

DETAILED DESCRIPTION:
This research was planned as a randomized controlled experimental type to determine the effect of playing with a toy nebulizer and watching cartoons on children's fear and physiological parameters in 3-6 year old children who were administered inhaler medication. The population of the study, planned as a randomized controlled experimental study, will consist of 4-6 year old children who apply to Tarsus State Hospital pediatric services and receive inhaler treatment. According to the power analysis performed for the sample size, the power of the sample was calculated with the G*Power 3.1 program, in line with the literature. While the amount of Type I error was 0.05 and the power of the test was 0.95 (α= 0.05, 1-β= 0.95), the minimal sample size was calculated as 105 children (35 children in each group). Considering the possible losses from the sample for any reason during the study period, it was planned to increase the number of samples by 10% and include 38 children in the study and control groups. Child Information Form, Fear Assessment Scale and Child Anxiety Scale-State Scale will be used to collect data.

Data collection In the study, children treated in pediatric emergency departments and administered inhaler medication will first be evaluated in terms of sampling criteria, and children who do not meet the criteria will be excluded from the study. The nurse researcher is the one who collects the data, evaluates it with the Fear and Anxiety Scale, and evaluates the physiological parameters.

Data analyses The data obtained in the study were analyzed using the Statistical Package for Social Sciences for Windows 25.0 program. Descriptive statistical methods (number, percentage, min-max values, mean and standard deviation) will be used when evaluating the data. The suitability of the data used to normal distribution will be checked with kurtosis and skewness values. In normally distributed data, when comparing quantitative data, an independent t-test will be used for the difference between two independent groups, and when comparing more than two dependent groups, analysis of variance will be applied in repeated measurements, and in case of a difference, Bonferroni will be used to find the group that makes the difference. In comparing quantitative data with non-normally distributed data, the Mann-Whitney U test will be applied for the difference between two independent groups, and in comparing more than two dependent groups, the Friedman test will be applied, and in case of a difference, the corrected Bonferroni will be used to find the group that makes the difference. Chi-square analysis will be applied to test the relationship between categorical variables. Cohen's Kappa Test will be applied in interobserver agreement analysis.

ELIGIBILITY:
Inclusion Criteria:

* The child is between 4 and 6 years old,
* No communication problems (visual/auditory/mental),
* Oxygen saturation is 90% or above,
* The child does not have a disease that may affect his/her life,
* Parent and child volunteering to participate in the research.

Exclusion Criteria:

* Nebul drug administration
* The child has visual, hearing, and mental disabilities,
* Having taken medication with a nebulizer before

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 114 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-11-19 (Actual); Study Completion 2024-11-19 (Actual)

PRIMARY OUTCOMES:
fear | 1 day
  Child Fear Scale is used to evaluate the anxiety/fear level of children. The scale uses cartoon faces consisting of five pictures and the anxiety/fear level is evaluated with numbers between "0" and "4". The first picture shows a score of "0", that is, "no anxiety/fear is felt", and the last picture shows a score of "4", that is, "the most severe anxiety/fear". As the score increases, the level of anxiety/fear also increases.
anxiety | 1 day
  Child Anxiety Scale-The State scale resembles a thermometer with a bulb at the bottom and horizontal lines at intervals going upwards. This scale, for children ages 4 to 10, asks children, "Imagine that all your anxious or nervous emotions are in the bulb or bottom part of the thermometer," or "If you are a little anxious or nervous, the emotions might move up a little bit on the thermometer." If you're very, very anxious or nervous, emotions can run rampant. "Put a line on the thermometer that shows how anxious or angry you are." To measure state anxiety, the child is asked to indicate what he or she is feeling "right now." The score can vary between 0-10.

CONTACTS AND LOCATIONS:
Locations (1):
- Tarsus State Hospital, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Conk, Z. Başbakkal, Z. Yılmaz, H. Bolışık, B. (2013). Pediatri Hemşireliği, Ankara:Akademisyen Tıp Kitabevi.
- [Background] Erdinç, E. (2022). Evde Nebülizatör Tedavisi Kime? Nasıl?. ToraksDergisi, 3(2), 21-25. Retrieved from https://turkthoracj.org/content/files/sayilar/93/buyuk/pdf_Toraksder_197.pdf
- [Background] Nilsson S, Finnstrom B, Kokinsky E, Enskar K. The use of Virtual Reality for needle-related procedural pain and distress in children and adolescents in a paediatric oncology unit. Eur J Oncol Nurs. 2009 Apr;13(2):102-9. doi: 10.1016/j.ejon.2009.01.003. Epub 2009 Feb 20. PMID 19230769
- [Background] Zengin M, Yayan EH, Duken ME. The Effects of a Therapeutic Play/Play Therapy Program on the Fear and Anxiety Levels of Hospitalized Children After Liver Transplantation. J Perianesth Nurs. 2021 Feb;36(1):81-85. doi: 10.1016/j.jopan.2020.07.006. Epub 2020 Nov 3. PMID 33158746
- [Background] Coskunturk AE, Gozen D. The Effect of Interactive Therapeutic Play Education Program on Anxiety Levels of Children Undergoing Cardiac Surgery and Their Mothers. J Perianesth Nurs. 2018 Dec;33(6):781-789. doi: 10.1016/j.jopan.2017.07.009. Epub 2018 Feb 3. PMID 29398304
- [Background] Durak H, Uysal G. The Effect of Cartoon Watching and Distraction Card on Physiologic Parameters and Fear Levels During Inhalation Therapy in Children: A Randomized Controlled Study. J Trop Pediatr. 2021 Jan 29;67(1):fmab018. doi: 10.1093/tropej/fmab018. PMID 33742204